CLINICAL TRIAL: NCT00424125
Title: Improving Pediatric Asthma Care in the District of Columbia (IMPACT DC)-Community Pharmacy Intervention
Brief Title: Involving Community Pharmacies in Improving Asthma Outcomes in an Urban Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen J. Teach, MD, MPH (Other)
Collaborators: National Association of Chain Drug Stores (Industry)
Responsible Party: Sponsor-Investigator, Stephen J. Teach, MD, MPH, Chief, Division of Allergy and Immunology, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IMPACT DC CPIT
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Asthma
Keywords: Asthma; Compliance; Randomized clinical trial
MeSH Terms: conditions — Asthma; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- Enhanced Pharmacy Care (Experimental): Received enhanced community pharmacy based services.
  Interventions: Behavioral: Enhanced Pharmacy Care; Behavioral: Control

INTERVENTIONS:
Behavioral: Enhanced Pharmacy Care — Participants randomized to "Enhanced Pharmacy Care" will have their prescriptions electronically transmitted or faxed to one of the five participating pharmacies.
  Pharmacists will then provide real-time, targeted education around the purpose and use of the new and refilled ICS medications to study participants and their families at each point of contact, including rationale for their use, device teaching, dosage review, and importance of compliance. Families randomized to "enhanced care" will also be contacted monthly by phone and mail with reminders to fill their controller medications prescriptions and to seek ongoing longitudinal asthma care with their primary care providers.
Behavioral: Control — Usual care.

SUMMARY:
This study seeks to determine whether education provided in community pharmacies and monthly reminder calls can improve compliance with asthma medications.

We hypothesize that those pediatric patients with asthma 12 months to 12 years of age who receive comprehensive asthma care as part of a validated intervention (1) who are randomized to receive enhanced community pharmacy care will have significantly greater compliance with inhaled corticosteroids (ICS) six months after enrollment when compared with patients receiving usual pharmacy care. As secondary outcomes, we further hypothesize that they will have less unscheduled healthcare utilization and improved functional outcomes and QOL.

(1) Teach SJ, Crain EF, Quint DM, Hylan ML, Joseph JG. Improved Asthma Outcomes in a High Morbidity Pediatric Population: Results of an Emergency Department-based Randomized Clinical Trial. Archives of Pediatric and Adolescent Medicine. 2006;160:535-541.

DETAILED DESCRIPTION:
IMPACT DC has been funded by the National Association of Chain Drug Stores Foundation (NACDSF) to undertake a project regarding coordination between the existing IMPACT DC Asthma Clinic and certain community pharmacies in Northwest, Northeast, and Southeast DC that provide patients with asthma medications, devices, and education.

This is a single blind prospective randomized clinical trial in which eligible patients with asthma aged 12m to 12y, inclusive, seen in the current IMPACT DC Asthma Clinic and prescribed ICS as controller medications is randomized to either "usual pharmacy care" or "enhanced pharmacy care." The IMPACT DC Asthma Clinic is an ED-based follow-up clinic that has been shown to improve outcomes. (1)

Outcomes will be assessed by blinded and structured patient phone interview at 1, 3, and 6 months.

Patients randomized to usual pharmacy care will fill prescriptions by their usual preferred method, whereas patients randomized to enhanced pharmacy care will have these same prescriptions electronically transmitted to specifically trained pharmacists at one of the participating community pharmacies. Both "usual pharmacy care" and "enhanced pharmacy care" will be provided within all participating pharmacy sites.

Community pharmacies located in five zip codes in Northeast and Southeast DC with the highest absolute numbers of pediatric ED asthma visits to hospital in the District (20019, 20020, 20032, 20002, 20011) will be selected for the program based on their geographic distribution and ability to meet programmatic expectations. Pharmacies will receive electronically transmitted, faxed or verbal prescriptions from the IMPACT DC Asthma Clinic staff for patients identified as study participants in the intervention group.

Pharmacists will then provide real-time, targeted education around the purpose and use of the new and refilled ICS medications to study participants and their families at each point of contact, including rationale for their use, device teaching, dosage review, and importance of compliance. Families randomized to "enhanced care" will also be contacted monthly by phone and mail with reminders to fill their controller medications prescriptions and to seek ongoing longitudinal asthma care with their primary care providers.

(1) Teach SJ, Crain EF, Quint DM, Hylan ML, Joseph JG. Improved Asthma Outcomes in a High Morbidity Pediatric Population: Results of an Emergency Department-based Randomized Clinical Trial. Archives of Pediatric and Adolescent Medicine. 2006;160:535-541.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include:

  1. age between 12 months and 12 years, inclusive;
  2. prior physician-diagnosed asthma;
  3. prescription of an inhaled corticosteroid during the IMPACT DC Asthma Clinic visit,
  4. a parent/guardian available for interview;
  5. residence in one of the 5 zip codes in Washington, DC with the highest absolute numbers for asthma visits to the Emergency Department at Childrens National Medical Center (20019, 20020, 20032, 20002, 20011), and
  6. insurance that covers at least part of the cost of medications.

Exclusion Criteria:

* Exclusion criteria include:

  1. significant medical co-morbidities affecting the cardiorespiratory system;
  2. enrollment in another asthma research study;
  3. unavailability for telephone follow-up; or
  4. primary language other than English.

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2006-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Compliance with inhaled corticosteroids | 6 months following enrollment

SECONDARY OUTCOMES:
Unscheduled healthcare utilization for asthma | 6 months following enrollment
Quality of Life | 6 months following enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Teach, MD, MPH, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Teach SJ, Crain EF, Quint DM, Hylan ML, Joseph JG. Improved asthma outcomes in a high-morbidity pediatric population: results of an emergency department-based randomized clinical trial. Arch Pediatr Adolesc Med. 2006 May;160(5):535-41. doi: 10.1001/archpedi.160.5.535. PMID 16651498